CLINICAL TRIAL: NCT00044980
Title: Fresh Start: Promoting Health in Prostate Cancer Survivors
Brief Title: Diet and Exercise-Based Counseling Program Compared With a Standard Counseling Program in Patients With Early-Stage Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Other
Other Study IDs: Pro00008521; DUMC-1306-04-7R3ER; DUMC-1306-01-7R2ER; NCI-H02-0090; CDR0000069500
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2012-11

CONDITIONS: Malnutrition; Prostate Cancer
Keywords: malnutrition; stage I prostate cancer; stage II B prostate cancer; stage II A prostate cancer
MeSH Terms: conditions — Malnutrition; Prostatic Neoplasms | interventions — Nutritional Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: nutritional support
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: An individualized, computer-designed health program may promote changes in diet and physical activity and may improve quality of life in patients who have early-stage prostate cancer.

PURPOSE: Randomized clinical trial to compare the effectiveness of an individualized, computer-designed diet and exercise-based counseling program with that of a standard counseling program in promoting health in patients who have early-stage prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effectiveness of a computer-tailored, correspondence course vs standardized materials in promoting changes in diet and physical activity (PA) behaviors in patients with early stage prostate or breast (closed to accrual as of 8/1/03) cancer who currently do not practice goal behavior in at least 2 of the following 3 areas: performance of moderate PA for at least 150 minutes per week; consumption of at least 5 servings of vegetables or fruit daily; or consumption of a diet with less than 30% fat (with less than 10% of kilocalories from either saturates or polyunsaturates).
* Compare the health and quality of life of patients treated with these interventions.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients participate in a computer-tailored, correspondence course comprising personalized diet and exercise intervention and other health information over a 10-month period.
* Arm II: Patients receive usual care comprising standardized print materials related to diet, exercise, cancer, and other pertinent health issues over a 10-month period.

In both arms, diet and exercise behavior, quality of life, co-morbidity status, depression, social support, worry, self efficacy, and coping style are assessed during phone interviews conducted at baseline, after completion of 10 months of study intervention, and then at 1 year. Intervention usefulness is assessed after completion of 10 months of study intervention.

Patients in both arms who live within a 1-hour drive from Duke University Medical Center may undergo blood draw to test for substances related to fruit and vegetable intake and measurement of height and weight. Patients may also be asked to wear a pedometer for a 1-week period.

PROJECTED ACCRUAL: A total of 530 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with early stage prostate or breast (closed to accrual as of 8/1/03) cancer within the past 9 months
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Breast cancer (closed to accrual as of 8/1/03) patients must be female

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No other malignancy within the past 5 years except nonmelanoma skin cancer
* Able to speak and write in English
* Performs insufficient exercise
* Maintains a high-fat, low-vegetable, low-fruit diet

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-07; Primary Completion 2005-09 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Demark-Wahnefried, PhD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Demark-Wahnefried W, Clipp EC, McBride C, Lobach DF, Lipkus I, Peterson B, Clutter Snyder D, Sloane R, Arbanas J, Kraus WE. Design of FRESH START: a randomized trial of exercise and diet among cancer survivors. Med Sci Sports Exerc. 2003 Mar;35(3):415-24. doi: 10.1249/01.MSS.0000053704.28156.0F. PMID 12618570
- [Background] Macri JM, Downs SM, Demark-Wahnefried W, Snyder DC, Lobach DF. A simple, flexible and scalable approach for generating tailored questionnaires and health education messages. Comput Inform Nurs. 2005 Nov-Dec;23(6):316-21. doi: 10.1097/00024665-200511000-00007. PMID 16292046
- [Result] Christy SM, Mosher CE, Sloane R, Snyder DC, Lobach DF, Demark-Wahnefried W. Long-term dietary outcomes of the FRESH START intervention for breast and prostate cancer survivors. J Am Diet Assoc. 2011 Dec;111(12):1844-51. doi: 10.1016/j.jada.2011.09.013. PMID 22117660
- [Result] Ottenbacher AJ, Day RS, Taylor WC, Sharma SV, Sloane R, Snyder DC, Kraus WE, Demark-Wahnefried W. Exercise among breast and prostate cancer survivors--what are their barriers? J Cancer Surviv. 2011 Dec;5(4):413-9. doi: 10.1007/s11764-011-0184-8. Epub 2011 May 20. PMID 21598023
- [Result] Demark-Wahnefried W, Clipp E, Lipkus I, et al.: Results of FRESH START: a randomized controlled trial to improve diet and exercise behaviors in breast and prostate cancer survivors. [Abstract] J Clin Oncol 24 (Suppl 18): A-8503, 468s, 2006.
- [Result] Demark-Wahnefried W, Clipp EC, Lipkus IM, Lobach D, Snyder DC, Sloane R, Peterson B, Macri JM, Rock CL, McBride CM, Kraus WE. Main outcomes of the FRESH START trial: a sequentially tailored, diet and exercise mailed print intervention among breast and prostate cancer survivors. J Clin Oncol. 2007 Jul 1;25(19):2709-18. doi: 10.1200/JCO.2007.10.7094. PMID 17602076
- [Result] Snyder DC, Sloane R, Lobach D, Lipkus I, Clipp E, Kraus WE, Demark-Wahnefried W; Fresh Start study. Agreement between a brief mailed screener and an in-depth telephone survey: observations from the Fresh Start study. J Am Diet Assoc. 2004 Oct;104(10):1593-6. doi: 10.1016/j.jada.2004.07.024. PMID 15389420
- [Result] Mosher CE, Lipkus IM, Sloane R, Kraus WE, Snyder DC, Peterson B, Jones LW, Demark-Wahnefried W. Cancer survivors' health worries and associations with lifestyle practices. J Health Psychol. 2008 Nov;13(8):1105-12. doi: 10.1177/1359105308095964. PMID 18987083
- [Result] Mosher CE, Fuemmeler BF, Sloane R, Kraus WE, Lobach DF, Snyder DC, Demark-Wahnefried W. Change in self-efficacy partially mediates the effects of the FRESH START intervention on cancer survivors' dietary outcomes. Psychooncology. 2008 Oct;17(10):1014-23. doi: 10.1002/pon.1327. PMID 18300337
- [Result] Snyder DC, Sloane R, Lobach D, Lipkus IM, Peterson B, Kraus W, Demark-Wahnefried W. Differences in baseline characteristics and outcomes at 1- and 2-year follow-up of cancer survivors accrued via self-referral versus cancer registry in the FRESH START Diet and exercise trial. Cancer Epidemiol Biomarkers Prev. 2008 May;17(5):1288-94. doi: 10.1158/1055-9965.EPI-07-0705. PMID 18483353
- [Result] Sloane R, Snyder DC, Demark-Wahnefried W, Lobach D, Kraus WE. Comparing the 7-day physical activity recall with a triaxial accelerometer for measuring time in exercise. Med Sci Sports Exerc. 2009 Jun;41(6):1334-40. doi: 10.1249/MSS.0b013e3181984fa8. PMID 19461530
- [Result] Mosher CE, Sloane R, Morey MC, Snyder DC, Cohen HJ, Miller PE, Demark-Wahnefried W. Associations between lifestyle factors and quality of life among older long-term breast, prostate, and colorectal cancer survivors. Cancer. 2009 Sep 1;115(17):4001-9. doi: 10.1002/cncr.24436. PMID 19637244
- [Result] Ottenbacher A, Sloane R, Snyder DC, Kraus W, Sprod L, Demark-Wahnefried W. Cancer-specific concerns and physical activity among recently diagnosed breast and prostate cancer survivors. Integr Cancer Ther. 2013 May;12(3):206-12. doi: 10.1177/1534735412449734. Epub 2012 Aug 9. PMID 22879576
- [Result] Mosher CE, Lipkus I, Sloane R, Snyder DC, Lobach DF, Demark-Wahnefried W. Long-term outcomes of the FRESH START trial: exploring the role of self-efficacy in cancer survivors' maintenance of dietary practices and physical activity. Psychooncology. 2013 Apr;22(4):876-85. doi: 10.1002/pon.3089. Epub 2012 Apr 30. PMID 22544562
- [Result] Ottenbacher AJ, Day RS, Taylor WC, Sharma SV, Sloane R, Snyder DC, Lipkus IM, Jones LW, Demark-Wahnefried W. Long-term physical activity outcomes of home-based lifestyle interventions among breast and prostate cancer survivors. Support Care Cancer. 2012 Oct;20(10):2483-9. doi: 10.1007/s00520-011-1370-y. Epub 2012 Jan 17. PMID 22249915
- [Result] Wilkinson AV, Barrera SL, McBride CM, Snyder DC, Sloane R, Meneses KM, Pekmezi D, Kraus WE, Demark-Wahnefried W. Extant health behaviors and uptake of standardized vs tailored health messages among cancer survivors enrolled in the FRESH START trial: a comparison of fighting-spirits vs fatalists. Psychooncology. 2012 Jan;21(1):108-13. doi: 10.1002/pon.1870. Epub 2010 Nov 8. PMID 21061408
- [Result] Demark-Wahnefried W. Print-to-Practice: Designing Tailored Print Materials to Improve Cancer Survivors' Dietary and Exercise Practices in the FRESH START Trial. Nutr Today. 2007 May;42(3):131-138. doi: 10.1097/01.NT.0000277790.03666.95. No abstract available. PMID 19081749
- [Result] Stull VB, Snyder DC, Demark-Wahnefried W. Lifestyle interventions in cancer survivors: designing programs that meet the needs of this vulnerable and growing population. J Nutr. 2007 Jan;137(1 Suppl):243S-248S. doi: 10.1093/jn/137.1.243S. PMID 17182834
- [Result] Adams RN, Mosher CE, Blair CK, Snyder DC, Sloane R, Demark-Wahnefried W. Cancer survivors' uptake and adherence in diet and exercise intervention trials: an integrative data analysis. Cancer. 2015 Jan 1;121(1):77-83. doi: 10.1002/cncr.28978. Epub 2014 Aug 25. PMID 25155573
- [Result] Morey MC, Blair CK, Sloane R, Cohen HJ, Snyder DC, Demark-Wahnefried W. Group trajectory analysis helps to identify older cancer survivors who benefit from distance-based lifestyle interventions. Cancer. 2015 Dec 15;121(24):4433-40. doi: 10.1002/cncr.29684. Epub 2015 Oct 29. PMID 26512712